CLINICAL TRIAL: NCT02994901
Title: Cause and Importance of the Age-dependent Sarcopenia With a Blood Based Bioenergetics & Cytokine Profiling Approach
Brief Title: Cause and Importance of the Age-dependent Sarcopenia
Acronym: SARCOPENIA
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Kristina Norman, PD Dr., Charite University, Berlin, Germany
Other Study IDs: EA1/260/16
Record Dates: First submitted 2016-12-07; First posted 2016-12-16 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Geriatrics; Biomarker
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Geriatric patient with Sarcopenia
- Group 2: Geriatric Patient without Sarcopenia
- Group 3: healthy control group

SUMMARY:
The goal of this cross-sectional study is to evaluate the difference in cytokine profiling approach and mitochondrial function between geriatric sarcopenic patients (group 1) and geriatric non-sarcopenic patients (group 2) and healthy (group 3) geriatric participants.

DETAILED DESCRIPTION:
Study participants (group 1&2) are assessed during the hospital stay and age-matched controls (group 3) will be recruited through Flyers.

The investigators aim to isolate and cryopreserve peripheral blood mononuclear cells (PBMCs) from whole blood to perform functional assays on mitochondrial respiratory capacity and ROS. Furthermore, the investigators will investigate the association between biomarkers and frailty, quality of life, functional performance, fatigue and risk of depression.

The investigators hypothesize that this profiling approach will allow the evaluation of the progression of age-dependent sarcopenia and uncover novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 85 years
* Informed written consent
* Normal cognitive status according to Mini-Mental State Examination (MMSE ≥ 24 points)
* Life expectancy of > 3 months according to treating doctor
* without implanted Defibrillation
* without acute Sepsis
* without neurodegenerative diseases, especially amyotrophic lateral sclerosis (ALS) and Huntington

Exclusion Criteria:

* Age < 60 years or > 85 years
* Lack of informed written consent
* Low cognitive status according to Mini-Mental State Examination (MMSE < 24 points)
* Life expectancy of < 3 months according to treating doctor
* Implanted Defibrillation
* Acute Sepsis
* neurodegenerative diseases, especially amyotrophic lateral sclerosis (ALS) and Huntington

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: sarcopenic patient Group 2: non-sarcopenic patient Group 3: healthy control
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Differences in mitochondrial respiratory capacity of peripheral blood mononuclear cells (PBMCs) using Oxygraph-2k respirometry | Baseline

SECONDARY OUTCOMES:
Quality of life (validated questionnaire) | Baseline
Frailty Status according to Fried et.al. criteria | Baseline
Functional limitations (single validated questionnaire) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Norman, PD Dr., Principal Investigator — Charite Research Group on Geriatrics
Locations (1):
- Charite University Medicine, Research Group on Geriatrics, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marzetti E, Calvani R, Cesari M, Buford TW, Lorenzi M, Behnke BJ, Leeuwenburgh C. Mitochondrial dysfunction and sarcopenia of aging: from signaling pathways to clinical trials. Int J Biochem Cell Biol. 2013 Oct;45(10):2288-301. doi: 10.1016/j.biocel.2013.06.024. Epub 2013 Jul 8. PMID 23845738
- [Background] Leger B, Derave W, De Bock K, Hespel P, Russell AP. Human sarcopenia reveals an increase in SOCS-3 and myostatin and a reduced efficiency of Akt phosphorylation. Rejuvenation Res. 2008 Feb;11(1):163-175B. doi: 10.1089/rej.2007.0588. PMID 18240972